CLINICAL TRIAL: NCT01144975
Title: A Randomized Study of the Safety and Biologic Activity of XOMA 052 in Subjects With Type 2 Diabetes Mellitus on Stable Metformin Monotherapy
Brief Title: Study of the Safety and Biologic Activity of XOMA 052 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X052118
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Type 2; Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- XOMA 052 (Active Comparator)
  Interventions: Drug: XOMA 052
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XOMA 052 — Sterile solution, dose level varies by dose group and study drug administration day, SC injections administered by study personnel at time points specified in the protocol (the subject will receive a total of 8 injections)
  Arms: XOMA 052
Drug: Placebo — Sterile solution, SC injections administered by study personnel (the subject will receive a total of 8 injections)
  Arms: Placebo

SUMMARY:
The study hypothesis is that XOMA 052 is likely to improve glycemic control in subjects with Type 2 Diabetes Mellitus.

The purpose of this study is to determine whether XOMA 052 improves glycemic control in subjects on Metformin monotherapy whose diabetes is still not adequately controlled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D (disease duration >= 6 months)
* HbA1c measurements >= 7.0% and <= 10.0%
* On a stable regimen of metformin monotherapy
* Age >= 18 and <= 75
* Stable diet and exercise regimen
* BMI <= 40 kg/m2

Exclusion Criteria:

* Significant signs and symptoms of uncontrolled hyperglycemia (i.e., polyuria, polydipsia, or polyphagia)
* Uncontrolled hypertension (systolic > 170 mmHg and/or diastolic > 110 mmHg)
* Known to be positive for Hep B surface antigen (HBsAg), Hep C virus (HCV), or HIV
* History of allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Advanced stage heart failure (New York Heart Association [NYHA] class 3 or 4)
* Pulmonary disease requiring medication other than inhaled corticosteroid s
* History of tuberculosis or positive PPD test.
* Active leg, foot, or decubitus ulcer
* Any significant inflammatory, rheumatologic, or systemic autoimmune disease
* History or any symptoms of a demyelinating disease
* History of severe non-proliferative or proliferative retinopathy

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety assessed by pre- and post-treatment serial measurements of vital signs, clinical laboratory assessments, daily fasting blood glucose measured by the subject using a glucose monitor, and treatment-emergent adverse events. | Day 0 pre-dose through Day 420

SECONDARY OUTCOMES:
Pharmacokinetic assessments of XOMA 052 from serum samples collected at time points specified in the protocol. | Day 0 pre-dose through Day 420
Anti-inflammatory activity measured by hs-CRP and cytokines collected at time points specified in the protocol. | Day 0 pre-dose through Day 420
Anti-diabetic activity measured by HbA1c, FPG, OGTT, C-peptide, and insulin collected at time points specified in the protocol. | Day 0 pre-dose through Day 420

CONTACTS AND LOCATIONS:
Locations (1):
- Mexico City, Mexico